CLINICAL TRIAL: NCT04558775
Title: Tran-epidermal Water Loss (TEWL) as a Predictive Marker for Diabetic Foot Ulcer (DFU) Recurrence
Brief Title: TEWL Biomarker Study for Diabetic Foot Ulcer Recurrence
Acronym: TEWL
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Indiana University (Other); Stanford University (Other); University of Miami (Other); University of Pittsburgh (Other); University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Cathie Spino, ScD, Research Professor of Biostatistics, SABER Director, University of Michigan
Other Study IDs: HUM00176334; 1U24DK122927-01 (NIH)
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Diabetes; Diabetic Foot; Diabetic Foot Ulcer; Diabetic Wound; Diabetic
Keywords: biomarker; TEWL; trans epidermal water loss; DFC; Diabetic Foot Consortium
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — no intervention

SUMMARY:
This is a multicenter study of patients with diabetic foot ulcers (DFU) to develop and validate potential tissue-based biomarkers that predict DFU wound recurrence. Trans-epidermal water loss (TEWL) will be measured on the closed wound site and a location similar to the wound site (reference site). Participants will be enrolled within two weeks after closure of their DFU. Complete wound healing will be verified at a second visit two weeks later and this visit will start the 16 week timeline where participants will be followed weekly by phone until the earliest of DFU wound recurrence or 16 weeks. Participants who experience a DFU wound recurrence and a subset of participants who do not experience a DFU wound recurrence by week 16 will be asked to attend one final visit.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria at Visit 1:

1. Age > 18 years.
2. Willing and able to comply with protocol instructions.
3. Clinically diagnosed DFU is closed.
4. Clinically diagnosed with diabetes or meeting the American Diabetes Association (ADA) criteria.
5. Provides written informed consent.

   At Visit 2, confirmation of complete wound healing, the following additional inclusion criterion must be met:
6. Confirmation that the target DFU that was assessed as healed at Visit 1 remains healed two weeks later (at Visit 2).

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. DFU wounds closed more than 2 weeks before Visit 1, or to be closed by flap or graft coverage
2. Closed DFU site whose size or location would not allow five separate TEWL measurements
3. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diabetic patients with diabetic foot ulcer
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who have DFU wound recurrence by 16 weeks after complete wound healing | 1 up to 16 weeks after wound closure

SECONDARY OUTCOMES:
Time to DFU wound recurrence after complete wound healing | Up to 16 weeks after wound closure
Participant self-report of DFU wound recurrence | 16 weeks
Clinician assessment of DFU wound recurrence | 16 weeks
  Concordance between participant self-report and clinician assessment of DFU wound recurrence is important to provide confidence in the use of patient-reports for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Study Chair — Indiana University
Locations (6):
- United States (6):
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided